CLINICAL TRIAL: NCT06156280
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, and Efficacy of TQH2929 in Healthy Adult Subjects
Brief Title: A Clinical Study of TQH2929 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQH2929-I-01 (Ia)
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TQH2929 Injection (1 mg/kg) (Experimental): TQH2929 Injection 1 mg/kg is administered as a single dose.
  Interventions: Drug: TQH2929 injection
- TQH2929 Injection (3 mg/kg) (Experimental): TQH2929 Injection 3 mg/kg is administered as a single dose.
  Interventions: Drug: TQH2929 injection
- TQH2929 Injection (10 mg/kg) (Experimental): TQH2929 Injection 10 mg/kg is administered as a single dose.
  Interventions: Drug: TQH2929 injection
- TQH2929 Injection (20 mg/kg) (Experimental): TQH2929 Injection 20 mg/kg is administered as a single dose.
  Interventions: Drug: TQH2929 injection
- TQH2929 Injection (30 mg/kg) (Experimental): TQH2929 Injection 30 mg/kg is administered as a single dose.
  Interventions: Drug: TQH2929 injection
- Placebo Injection (Placebo Comparator): Placebo injection is administered as a single dose or multiple doses (once every two weeks).
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: TQH2929 injection — TQH2929 injection is a humanized monoclonal antibody that interfering with the signal cascade.
  Arms: TQH2929 Injection (1 mg/kg); TQH2929 Injection (10 mg/kg); TQH2929 Injection (20 mg/kg); TQH2929 Injection (3 mg/kg); TQH2929 Injection (30 mg/kg)
Drug: Placebo injection — Placebo comparator
  Arms: Placebo Injection

SUMMARY:
This project is divided into a single dose escalation and a multiple dose escalation phase Ia clinical study. This is a single-center, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetic characteristics of TQH2929 injection in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 55 years old (inclusive), both male and female;
* The male subject should weigh at least 50 kg, the female subject should weigh at least 45kg. And body mass index (BMI) within 19~26 kg/m2.
* Good health is defined as having no clinically relevant abnormalities identified by a detailed medical history, clinical signs, vital signs, full physical examination, 12-lead Electrocardiogram (ECG), Chest radiograph, abdominal ultrasound and clinical laboratory tests.
* Subjects voluntarily joined the study, sign informed consent form before the study and fully understand the study content.
* Have no pregnancy plan and voluntarily take effective contraception measures from time of screening to at least 6 months after the last dose (subjects and their partners).

Exclusion Criteria:

* Pregnant or lactating women;
* Past medical history or current cardiac, endocrine, metabolic, renal, hepatic, gastrointestinal, skin, infection, hematological, neurological or psychiatric diseases/abnormalities, or related chronic abnormalities, or related chronic diseases, or acute diseases, and evaluated the investigator to be not suitable for the trial;
* People who have abnormal and clinically significant results in vital signs, physical examination, laboratory tests, 12-lead ECG, Chest radiograph and abdominal ultrasound during screening period;
* Subjects positive for any of Hepatitis B Virus Surface Antigen (HBsAg), Hepatitis C Virus Antibody (Anti-HCV), Human Immunodeficiency Virus Antibody (Anti-HIV), and Treponema Pallidum Antibody (Anti-TP) tests;
* Subjects positive for tuberculoses spot (T-SPOT) result;
* Clinically significant infection requiring antibiotic or antiviral therapy prior to screening and the entire study period;
* Had undergone surgery within 4 weeks prior to screening period or expected to undergo surgery during the study period;
* Participated in any clinical trial within 3 months prior to the screening period;
* Received immunoglobulins or blood products within 30 days prior to randomization;
* Blood donation or significant blood loss of more than 400 mL within 2 months prior to randomization;
* People who have potential difficulty in blood collection, or have a history of needles or blood sickness；
* Any clear history of drug or food allergies, particularly those with allergies to similar components to the investigational drugs in this trial;
* People who have received or are planning to receive inactivated or active vaccines during the 30 days prior to randomization and the entire study period (including the follow-up period);
* Smoking more than 5 cigarettes per day or using equivalent amounts of nicotine or nicotine-containing products within 6 months prior to randomization, or those who cannot stop using any tobacco-based products during the trial;
* People who had long-standing alcohol abuse or alcohol consumption of more than 14 units (1 unit = 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) of alcohol per week within 3 months prior to screening, or those who cannot refrain from alcohol during the trial, or those who tested positive for alcohol breath;
* History of drug abuse or a positive result of urine drug test at screening;
* Received any marketed or investigational biologics within 4 months or 5 half-lives (whichever is longer) prior to randomization;
* Had taken any prescription drugs, over-the-counter drugs, or herbs within 4 weeks prior to randomization, with the exception of vitamin products;
* Use of any systemic cytotoxicity or systemic immunosuppressants within 6 months prior to randomization or during the study period, or any local cytotoxin or local immunosuppressive drug within 30 days or 5 half-life periods (whichever is longer) prior to randomization or during the study period;
* Any situation in which the investigator believes that this poses a safety risk to the subject in the trial or may interfere with the conduct of the study, or that the investigator believes that the subject may not be able to complete the study or may not be able to comply with the requirements of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE) rate | Single dose: Up to Day 113
  The occurrence of all adverse events (AE).
Serious adverse events (SAE) rate | Single dose: Up to Day 113
  The occurrence of all adverse events (SAE).
Treatment-related adverse events (TRAE) rate | Single dose: Up to Day 113
  The occurrence of all treatment-related adverse events (TRAE).
Incidence of clinical laboratory abnormalities | Single administration dose (SAD) group: up to Day 113
  Proportion of subjects with clinical laboratory abnormalities

SECONDARY OUTCOMES:
Time to reach maximum observed serum concentration (Tmax), SAD | 1 hour pre-dose, 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours postdose.
  Time to reach maximum (peak) serum concentration after administration in SAD group
Maximum serum concentration (Cmax), SAD | 1 hour pre-dose, 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours postdose.
  The maximum observed serum concentration of study drug in SAD group.
Area under the concentration-time curve from zero to infinity (AUC 0-∞), SAD | 1 hour pre-dose, 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours postdose.
  Area under the concentration-time curve of the TQH2929 Injection in serum over the time interval from 0 extrapolated to infinity in SAD group.
Area under the concentration-time curve from 0 to last observation (AUC 0-t), SAD | 1 hour pre-dose, 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours postdose.
  Area under the concentration-time curve of the TQH2929 Injection in serum over the time interval from 0 extrapolated to the last quantifiable data time-point in SAD group.
Apparent volume of distribution (Vd/F), SAD | 1 hour pre-dose, 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours postdose.
  Apparent volume of distribution of the TQH2929 Injection in serum in SAD group.
Apparent clearance (CL/F), SAD | 1 hour pre-dose, 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours postdose.
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body, in SAD group.
Half-life (t1/2), SAD | 1 hour pre-dose, 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours postdose.
  The time required for half of the drug to be eliminated from the serum in SAD group.
Anti-drug antibodies (ADA) | SAD group: 1 hour pre-dose, postdose on Day 15, Day 57, Day 85, Day 113.
  Proportion of subjects with a positive ADA reading at any time point during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China